CLINICAL TRIAL: NCT05337865
Title: Assessment of the Aerobic Capacity of (Well-trained) Transgender Women Athletes Submitted to the Maximal Exercise Test: a Prospective Cohort.
Brief Title: Transgender Observational Performance
Acronym: TOP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Leonardo Alvares, Medical Technical Director, Instituto Brasileiro de Controle do Cancer
Other Study IDs: 52428321.2.0000.0062
Record Dates: First submitted 2022-03-17; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Transgender Persons
Keywords: Transgender women; Oxygen uptake; Cardiac output; Muscle strength; Acute physical effort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Transgender women: Well-trained transgender women.
  Interventions: Other: Aerobic exercise test.
- Cisgender Women: Well-trained cisgender women.
  Interventions: Other: Aerobic exercise test.
- Cisgender Men: Well-trained cisgender men.
  Interventions: Other: Aerobic exercise test.

INTERVENTIONS:
Other: Aerobic exercise test. — Aerobic exercise test at a treadmill.

SUMMARY:
The study will evaluate the sports capabilities of transgender women mainly in terms of muscular strength and aerobic capacity (VO2max). The control group will be composed of cisgender women and cisgender men with the same levels of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a transgender woman by the DSM-V or ICD10.
* Gonadectomized and non-gonadectomized
* Initiation of androgen blockade and/or estrogen use after 12 years of age.
* Age range 18 to 50 years old.
* BMI: 18.0 to 34.9 kg/m2.
* Well-trained individuals (IPAQ very active)

Exclusion Criteria:

* Current or previous morbidities that could interfere with strength or aerobic tests.
* Chronic illnesses and/or chronic medication use.
* Musculoskeletal limitations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Well-trained Transgender women, cisgender men and cisgender women.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity change of transgender women over 12 months assessed by cardiopulmonary exercise testing (K5 - COSMED, Italia) on a treadmill (MOVEMENT/ET20 RT250G2SAC110V ) with incremental effort until exhaustion (ramp protocol). | Baseline, 6 months, 12 months after starting the observational study.
  The comparison of changes in aerobic capacity of transgender women, cigender women and cisgender men submitted to maximum effort Participants will be submitted to cardiopulmonary exercise testing (K5 - COSMED, Italia) on a treadmill (MOVEMENT/ET20 RT250G2SAC110V ) with incremental effort until exhaustion (ramp protocol). The maximum functional capacity will be determined by peak oxygen consumption (VO2peak) evaluated at the maximum exercise intensity.

SECONDARY OUTCOMES:
Skeletal muscle mass change of transgender women over 12 months assessed by a densitometry device (GE Prodigy). | Baseline, 6 months, 12 months after starting the observational study.
  The comparison of changes in skeletal muscle mass (kg) of transgender women, cisgender women and cisgender men over 12 months. Muscle mass will be assessed by a densitometry device (GE Prodigy) with X-ray absorptiometry technique with two whole-body energy levels and analyzed in the corresponding manufacturer's software.
Muscle strength change of transgender women over 12 months assessed by hand grip strength (HGS) test using the Jamar Hand Dynamometer | Baseline, 6 months, 12 months after starting the observational study.
  The comparison of changes in muscle strength of transgender women, cisgender women and cisgender men over 12 months. The hand grip strength (HGS) test will be carried out using the Jamar Hand Dynamometer by technique recommended by the American Society of Hand Therapists (ASHT) The tests will be performed with the dominant and non-dominant hands of each individual three consecutive times. Participants will be instructed to perform a maximum contraction for 3 seconds in each test. There will be a 30-second rest period between each test. To analyse the parameters associated with the measurement of HGS in each individual, the mean values (kg) of the three tests for each hand will be used according to the ASHT reference and considered the most reliable way to measure HGS. The maximum strength (kg) of each individual will be also analysed.
Vertical jump height changes of transgender women over 12 months assessed by the jumping mat (Elite Jump®, S2 Sports, São Paulo, Brazil) | Baseline, 6 months, 12 months after starting the observational study.
  The comparison of changes in vertical jump during sprint of transgender women, cisgender women and cisgender men over 12 months.Vertical jump heights (cm) will be evaluated using two different techniques - the jump with a static start at 90° of knee flexion for ~2s before the jump, and another free jump to make the descent movement and vertical impulse with leg extension. The depth of the countermovement will be determined by the participant himself, in order to avoid alterations in the coordination of the jump.
  All jumps must be performed with hands on hips and participants will be instructed to jump as high as possible.
  The jumping mat (Elite Jump®, S2 Sports, São Paulo, Brazil) will be used. A total of five attempts will be allowed for each jump, spaced by 15 second intervals. The highest height for each modality will be used for future analyses.
Speed changes of transgender women over 12 months assessed by 20-meter run with change of direction (Zig-Zag Test). | Baseline, 6 months, 12 months after starting the observational study.
  The comparison of changes of speed during sprint of transgender women, cisgender women and cisgender men over 12 months.Participants will be instructed to fast for at least 2 hours before the test, following the dietary recommendations described for the maximal effort test. Before the start of the tests, participants will be asked to perform a warm-up protocol including running for 10 minutes of light to moderate intensity, followed by 3 minutes of active lower limb stretching.
  We will use the 20-meter run with change of direction (Zig-Zag Test). There will be 3 changes of direction with cones at 100° of angulation. The average duration of execution of this test by trained individuals ranges between 5 and 6 seconds.
  Photocells will be used to start and stop the timer, in order to increase the accuracy of the test.
  Participants will take the test in 3 attempts, with a 15-minute break between them, for equipment adjustments and rest.
Heart rate change of transgender women over 12 months assessed by frequency meter (Polar®) during cardiopulmonary exercise testing | Baseline, 6 months, 12 months after starting the observational study.
  The comparison of changes in heart rate capacity of transgender women, cigender women and cisgender men submitted to maximum effort Participants will be submitted to cardiopulmonary exercise testing (K5 - COSMED, Italia) on a treadmill (MOVEMENT/ET20 RT250G2SAC110V ) with incremental effort until exhaustion (ramp protocol. Heart rate will be continuously evaluated through frequency meter (Polar®).
Percentage of body fat mass (%FM) change of transgender women over 12 months assessed by a densitometry device (GE Prodigy). | Baseline, 6 months, 12 months after starting the observational study.
  The comparison of changes in percentage of body fat mass (%FM), of transgender women, cisgender women and cisgender men over 12 months. Muscle mass will be assessed by a densitometry device (GE Prodigy) with X-ray absorptiometry technique with two whole-body energy levels and analyzed in the corresponding manufacturer's software.

IPD SHARING:
Plan to Share IPD: No
No sharing will be done.